CLINICAL TRIAL: NCT04980079
Title: Primary Versus Deferred Ureteroscopy for Management of Calculus Anuria in Children: A Prospective Randomized Study
Brief Title: Primary Versus Deferred Ureteroscopy for Calculus Anuria in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Mostafa, Principal Investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: calculus anuria in children
Record Dates: First submitted 2021-07-14; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Ureter Obstruction
MeSH Terms: conditions — Ureteral Obstruction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A -undergo primary ureteroscopy URS (Active Comparator): Thirty children with calicular anuria will undergo primary ureteroscopy URS
  Interventions: Procedure: Primary ureterscopy URS
- the group B(30 patients) will undergo deferred ureteroscopy URS (Active Comparator): group B (30) patients will be admitted to do urinary drainage through the insertion of a double-J stent or percutaneous nephrostomy (PCN) at first , then a deferred ureteroscopy URS will be done
  Interventions: Procedure: deferred ureteroscopy URS

INTERVENTIONS:
Procedure: Primary ureterscopy URS — Ureteral dilatation will be done when the stone size exceeds 10 mm to facilitate the extraction of the fragments. Ureteroscopic lithotripsy will be done using a 6.5:7.5 Fr semi-rigid ureteroscope and holmium laser. The ureteric stent will last for one week after lithotripsy
  Other Names: URSureteroscopy
  Arms: group A -undergo primary ureteroscopy URS
Procedure: deferred ureteroscopy URS — insertion of a double -J stent or percutaneous nephrostomy (PCN) at first , then a deferred ureteroscopy URS will be done .
  Arms: the group B(30 patients) will undergo deferred ureteroscopy URS

SUMMARY:
To evaluate the role of both primary and deferred URS in the management of calculus anuria concerning the feasibility, clinical outcome, and cost-effectiveness in children in a comparative study

DETAILED DESCRIPTION:
Thirty group B (30) patients will be admitted to do urinary drainage through the insertion of a JJ stent or percutaneous nephrostomy (PCN) at first , then a deferred URS will be done children will undergo primary URS( group A ) and in. Ureteral dilatation will be done when the stone size exceeds 10 mm to facilitate the extraction of the fragments. Ureteroscopic lithotripsy will be done using a 6.5:7.5 Fr semi-rigid ureteroscope and holmium laser. The ureteric stent will last for one week after lithotripsy. Postoperatively, the patients in both groups will monitored for post obstructive diuresis, fever, hematuria, and extent of renal function improvement.

ELIGIBILITY:
Inclusion Criteria:

* Children ˂12 years with calculus anuria.
* Clinically stable (serum creatinine < 3.5 mg/dl, blood urea < 100 mg/dl,serum potassium level < 7 milliequivalent /L and /or ph of blood > 7.1)
* All the patients free of sepsis.

Exclusion Criteria:

* Unstable children (serum creatinine ≥ 3.5 mg/dl, blood urea ≥ 100 mg/dl, serum potassium ≥ 7 milliequivalent/l, and/or blood pH ≤ 7.1, signs of acidosis, sepsis, or fluid retention).
* Children with underlying urological structural abnormalities

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-11-15 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
renal function | one month .
  improvement in creatinine level mg/dl urea level mg/dl

SECONDARY OUTCOMES:
the stone-free rates | one month
  The clinical outcomes of the procedures including the perioperative complications :
  * of perforation
  * of infection
  * of residual stones
  * of the stone-free rates

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa abdelrazek, MD, Study Director — SVU
Locations (1):
- Mostafa, Luxor, Egypt

IPD SHARING:
Plan to Share IPD: No